CLINICAL TRIAL: NCT06573996
Title: The Effect of Intraoral Transcutaneous Electrical Nerve Stimulation (TENS) on Pain Perception During Orthodontic Alignment and Leveling: a Randomized Clinical Trial
Brief Title: The Effect of Intraoral Transcutaneous Electrical Nerve Stimulation in Orthodontics Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Pacific (Other)
Responsible Party: Principal Investigator, Jonas Bianchi, Assistant Professor, University of the Pacific
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB2024-212
Record Dates: First submitted 2024-08-20; First posted 2024-08-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Orthodontic Appliance; Pain; Transcutaneous Electric Nerve Stimulation; Orthodontic Appliance Complication
Keywords: Orthodontic Pain; TENS Therapy; Orthodontic Alignment; Randomized Clinical Trial; Transcutaneous Electrical Nerve Stimulation (TENS); Dental Pain Eraser
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: This study employs a split-mouth, parallel design, where each participant serves as their own control. The active treatment (TENS device) is applied to one side of the mouth, while a placebo (non-functioning device) is applied to the other side, both during the same session. The allocation of sides (left or right) for the active treatment versus placebo is randomized. This design allows for direct intra-subject comparison of pain levels between the treated and untreated sides, minimizing variability in pain perception and enhancing the reliability of the study outcomes.
  Each arm represents one of the four possible treatment locations where either the TENS device or the placebo will be applied: upper right, upper left, lower right, and lower left.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Upper Right Side - Active TENS Device (Experimental): Participants will receive the active TENS device on the upper right side of their mouth. This arm is designed to evaluate the effectiveness of the TENS device in reducing pain during orthodontic alignment on this specific side of the upper arch.
  Interventions: Device: Active TENS Device
- Arm 2: Upper Left Side - Placebo/Sham Device (Sham Comparator): Participants will receive a placebo (non-functioning) device on the upper left side of their mouth. This arm serves as a control to compare pain levels with the side receiving the active TENS device.
  Interventions: Device: Intervention 2: Placebo/Sham Device
- Arm 3: Lower Right Side - Active TENS Device (Experimental): Participants will receive the active TENS device on the lower right side of their mouth. This arm is intended to assess the effectiveness of the TENS device in reducing pain during orthodontic alignment on this specific side of the lower arch.
  Interventions: Device: Active TENS Device
- Arm 4: Lower Left Side - Placebo/Sham Device (Sham Comparator): Participants will receive a placebo (non-functioning) device on the lower left side of their mouth. This arm also serves as a control, providing a basis for comparison with the side receiving the active TENS device.
  Interventions: Device: Intervention 2: Placebo/Sham Device

INTERVENTIONS:
Device: Active TENS Device — Description: The active TENS device, specifically the Dental Pain Eraser (DPE), is applied to the gums for about 2.5 minutes. This intervention is designed to modulate nerve activity to reduce pain during orthodontic alignment and leveling.
  Arms Associated:
  Arm 1: Upper Right Side - Active TENS Device Arm 3: Lower Right Side - Active TENS Device
  Arms: Arm 3: Lower Right Side - Active TENS Device; Upper Right Side - Active TENS Device
Device: Intervention 2: Placebo/Sham Device — The placebo/sham device is identical in appearance to the TENS device but does not deliver electrical stimulation. It is applied to the gums for 2.5 minutes to serve as a control.
  Arms Associated:
  Arm 2: Upper Left Side - Placebo/Sham Device Arm 4: Lower Left Side - Placebo/Sham Device
  Arms: Arm 2: Upper Left Side - Placebo/Sham Device; Arm 4: Lower Left Side - Placebo/Sham Device

SUMMARY:
The goal of this clinical trial is to determine whether an intraoral Transcutaneous Electrical Nerve Stimulation (TENS) device can reduce pain during orthodontic alignment and leveling in adolescents and adults. The study aims to compare the effectiveness of the TENS device in reducing pain on one side of the mouth, where the device is used, to the other side, where a non-functioning (placebo) device is applied.

The primary questions this study aims to answer are:

Does the TENS device effectively reduce pain during orthodontic treatment compared to the placebo? How do patients pain levels differ between the treated and untreated sides of the mouth?

Participants will:

Have an orthodontic appliance placed on their teeth. Experience the TENS device being applied to one side of their mouth for 2.5 minutes immediately after the appliance placement (brackets and wires).

Report their pain levels at various intervals after the procedure (immediately, 2 hours, 6 hours, 12 hours, 24 hours, 48 hours, and 72 hours).

This study includes up to 150 participants who are undergoing routine orthodontic treatment. The findings will help researchers understand whether the TENS device can effectively reduce discomfort during orthodontic procedures, potentially leading to better patient care and comfort.

DETAILED DESCRIPTION:
This randomized, triple-blind, split-mouth clinical trial investigates the efficacy of an intraoral Transcutaneous Electrical Nerve Stimulation (TENS) device in reducing pain during orthodontic alignment and leveling. The TENS device, specifically the Dental Pain Eraser (DPE), is designed to modulate nerve activity through neuromodulation, offering a non-pharmacologic method of pain relief.

Participants in the study will undergo standard orthodontic treatment involving the placement of full fixed appliances. Immediately after placing these appliances, the TENS device will be applied to the gums on one side of the mouth for 2.5 minutes, while a placebo device (non-functioning) will be applied to the other side. The assignment of sides will be randomized to minimize bias.

Study Design:

This study is a randomized, quadruple-blind, split-mouth clinical trial designed to evaluate the effectiveness of the intraoral Transcutaneous Electrical Nerve Stimulation (TENS) device, the Dental Pain Eraser (DPE), in reducing pain during orthodontic alignment and leveling. The trial will involve up to 150 participants, both adolescents and adults, undergoing routine orthodontic treatment.

Blinding:

The study is quadruple-blind, meaning that the investigator, participants, the clinicians applying the treatment, and the researchers analyzing the data will be unaware of which side of the mouth received the functioning TENS device versus the placebo. This blinding is critical to eliminating bias in the treatment, assessment, and analysis phases of the study.

Randomization:

Participants will be randomized to receive the TENS device on either the left or right side of their mouth, with the opposite side receiving a placebo (non-functioning) device. Randomization will be conducted using a computer-generated sequence to ensure an equal allocation of treatment across the study population.

Intervention:

TENS Device Application: The TENS device will be applied to the gums on one side of the mouth for 2.5 minutes immediately after the placement of full fixed orthodontic appliances.

Placebo Application: A placebo device that mimics the appearance and application of the TENS device but does not deliver electrical stimulation will be applied to the opposite side of the mouth for the same duration.

Pain Assessment:

Pain levels will be assessed using a Numeric Rating Scale (NRS) ranging from 0 (no pain) to 10 (worst pain imaginable). Assessments will be conducted at the following time points:

Immediately after appliance placement (0 hours) 2 hours post-placement 6 hours post-placement 12 hours post-placement 24 hours post-placement 48 hours post-placement 72 hours post-placement Participants will self-report their pain levels through a standardized survey administered via Google Forms. The survey will be designed to capture both the intensity and duration of pain experienced on each side of the mouth.

Data Collection and Management:

Data will be collected electronically and stored securely with password protection. Each participant's data will be de-identified, and only authorized research personnel will have access to the raw data. Pain ratings will be compiled into a spreadsheet for analysis, with data entry monitored to ensure accuracy.

Statistical Analysis:

The primary analysis will compare the pain levels between the side treated with the functioning TENS device and the placebo side. Paired t-tests will be used to assess the significance of any differences in pain levels. Secondary analyses may include subgroup analyses based on age, gender, and other demographic factors. The level of significance will be set at 0.05.

Detailed Description:

This randomized, triple-blind, split-mouth clinical trial investigates the efficacy of the Dental Pain Eraser (DPE), an intraoral Transcutaneous Electrical Nerve Stimulation (TENS) device, in reducing pain associated with orthodontic alignment and leveling. The DPE device is designed to provide a non-pharmacologic method of pain relief by modulating nerve activity through neuromodulation.

The trial involves up to 150 participants, including adolescents and adults, who are undergoing routine orthodontic treatment with full fixed appliances. The study's split-mouth design allows for intra-subject comparisons, enabling a direct assessment of the TENS device's effectiveness in pain management.

Participants will be randomly assigned to receive the TENS device on one side of their mouth, with the opposite side receiving a placebo device. Both the TENS and placebo devices will be applied for 2.5 minutes immediately after the placement of orthodontic appliances. The study is quadruple-blind, ensuring that neither the investigator, participants, clinicians, nor statisticians know which side received the active treatment.

Pain levels will be measured using a Numeric Rating Scale (NRS) at multiple time points following the orthodontic procedure. The primary outcome measure is the difference in pain levels between the treated and untreated sides of the mouth. Data will be collected via electronic surveys and analyzed using paired t-tests to determine the significance of any differences observed.

The results of this trial are expected to provide valuable insights into non-pharmacologic pain management strategies in orthodontics, potentially leading to improved patient outcomes and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

General Health: Patients who are generally healthy.

Orthodontic Treatment: Patients undergoing orthodontic treatment that requires the use of full-fixed appliances.

No Pain Medication: Patients not currently taking any medications for pain management.

Exclusion Criteria:

Patients with a history of seizures

Patients with or with a history of cardiac arrhythmias or pacemaker treatment

Patients taking any over-the-counter or prescription pain medication during the testing period.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-09-16 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Outcome Measure: Difference in Pain Levels Between Active TENS and Placebo | Pain will be measured at the following time points: immediately after appliance placement (0 hours), 2 hours, 6 hours, 12 hours, 24 hours, 48 hours, and 72 hours post-placement.
  The primary outcome measure is the difference in pain levels between the side of the mouth treated with the active TENS device and the side treated with the placebo device. Pain levels will be assessed using a Numeric Rating Scale (NRS) ranging from 0 (no pain) to 10 (worst pain imaginable).

SECONDARY OUTCOMES:
Duration of Pain Relief | Continuously measured from the time of appliance placement up to 72 hours post-placement.
  This outcome measure will compare the duration of pain relief provided by the intraoral TENS device versus the placebo. Participants will report when they first notice a reduction in pain and how long the relief lasts on each side of their mouth. The duration of pain relief will be recorded from the time of orthodontic appliance placement until the return of discomfort or pain.

CONTACTS AND LOCATIONS:
Locations (1):
- University of the Pacific, Arthur A. Dugoni School of Dentistry, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share individual participant data (IPD) is currently under consideration. The primary concerns include ensuring the privacy and confidentiality of participant data, as well as adhering to ethical guidelines and institutional policies. Additionally, the research team is evaluating the feasibility of de-identifying the data in a manner that protects participant identities while still providing valuable insights for future research. A final decision will be made based on these considerations, and the plan will be updated accordingly.

REFERENCES:
- [Background] Ngan P, Kess B, Wilson S. Perception of discomfort by patients undergoing orthodontic treatment. Am J Orthod Dentofacial Orthop. 1989 Jul;96(1):47-53. doi: 10.1016/0889-5406(89)90228-x. PMID 2750720
- [Background] Krishnan V. Orthodontic pain: from causes to management--a review. Eur J Orthod. 2007 Apr;29(2):170-9. doi: 10.1093/ejo/cjl081. PMID 17488999
- [Background] Inauen DS, Papadopoulou AK, Eliades T, Papageorgiou SN. Pain profile during orthodontic levelling and alignment with fixed appliances reported in randomized trials: a systematic review with meta-analyses. Clin Oral Investig. 2023 May;27(5):1851-1868. doi: 10.1007/s00784-023-04931-5. Epub 2023 Mar 6. PMID 36879148
- [Background] Sergl HG, Klages U, Zentner A. Pain and discomfort during orthodontic treatment: causative factors and effects on compliance. Am J Orthod Dentofacial Orthop. 1998 Dec;114(6):684-91. doi: 10.1016/s0889-5406(98)70201-x. PMID 9844209
- [Background] Brown DF, Moerenhout RG. The pain experience and psychological adjustment to orthodontic treatment of preadolescents, adolescents, and adults. Am J Orthod Dentofacial Orthop. 1991 Oct;100(4):349-56. doi: 10.1016/0889-5406(91)70073-6. PMID 1927986
- [Background] Roth PM, Thrash WJ. Effect of transcutaneous electrical nerve stimulation for controlling pain associated with orthodontic tooth movement. Am J Orthod Dentofacial Orthop. 1986 Aug;90(2):132-8. doi: 10.1016/0889-5406(86)90045-4. PMID 3488674
- [Background] Baghdadi ZD. Evaluation of electronic dental anesthesia in children. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1999 Oct;88(4):418-23. doi: 10.1016/s1079-2104(99)70055-7. PMID 10519748
- [Background] teDuits E, Goepferd S, Donly K, Pinkham J, Jakobsen J. The effectiveness of electronic dental anesthesia in children. Pediatr Dent. 1993 May-Jun;15(3):191-6. PMID 8378157
- [Background] Oztas N, Olmez A, Yel B. Clinical evaluation of transcutaneous electronic nerve stimulation for pain control during tooth preparation. Quintessence Int. 1997 Sep;28(9):603-8. PMID 9477875
- [Background] Haralambidis C. Pain-Free Orthodontic Treatment with the Dental Pain Eraser. J Clin Orthod. 2019 Apr;53(4):234-242. No abstract available. PMID 31390610
- [Background] Celebi F, Turk T, Bicakci AA. Effects of low-level laser therapy and mechanical vibration on orthodontic pain caused by initial archwire. Am J Orthod Dentofacial Orthop. 2019 Jul;156(1):87-93. doi: 10.1016/j.ajodo.2018.08.021. PMID 31256846